CLINICAL TRIAL: NCT05135364
Title: Hepatic Artery Infusion Chemotherapy (HAIC) Combined With Camrelizumab and Tyrosine Kinase Inhibitor for Unresectable Hepatocellular Carcinoma After Transcatheter Arterial Chemoembolization (TACE) Failure: a Single-arm and Open-label Prospective Study
Brief Title: HAIC Combined With Camrelizumab and TKI for Unresectable Hepatocellular Carcinoma After TACE Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yue Han (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yue Han, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3153
Record Dates: First submitted 2021-10-26; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Unresectable; TACE Failure; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+HAIC+TKI* (Experimental): *For patients who have not received molecular targeted therapy in the past, lenvatinib is recommended; For patients who have received sorafenib or lenvatinib in the past, regorafenib is recommended.
  Interventions: Drug: Camrelizumab; Drug: HAIC; Drug: TKI

INTERVENTIONS:
Drug: Camrelizumab — Each infusion is 30 min (not less than 20 min, not more than 60 min), once every 3 weeks
Drug: HAIC — A chemotherapy regimen perfused through the tumor supplying artery, d1-2 administration, perfused every 4 weeks
Drug: TKI — Lenvatinib or Regorafenib

SUMMARY:
The efficacy and safety of HAIC combined with tyrosine kinase inhibitor and immunotherapy have been proved by the clinical research. In this single-arm, open-label, prospective study, for those patients with unresectable primary HCC, in the case of failure of TACE treatment, the combination of HAIC, TKI and immunotherapy is expected to bring new breakthroughs.

ELIGIBILITY:
Inclusion Criteria:

1. Paticipants voluntarily joined the study and signed the informed consent form
2. Above 18 years old, both male and female
3. Clinical diagnosis or histopathologically confirmed advanced hepatocellular carcinoma (unresectable)
4. Child-Pugh score ≤ 7
5. BCLC B and C
6. TACE failure: ① Even if chemotherapeutic drugs are changed or the blood supply artery is reassessed, CT/MRI examinations after 2 consecutive TACE treatments 1-3 months show that the target lesions in the liver are compared with the previous TACE count. There are still more than 50% remaining or new lesions; ② extrahepatic metastasis or vascular invasion; ③ postoperative tumor indicators continue to rise (even if there is a short-term decline)
7. ECOG 0-1
8. The expected survival is more than 3 months
9. The function of vital organs is normal (no blood components, cell growth factor drugs are allowed to be used within 14 days before the first medication)
10. Women of childbearing age need contraception

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease
2. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other curative hormones), and continues to use it within 2 weeks before enrollment
3. Patients who have progressed after receiving second-line or above anti-vascular drug therapy in the past, or patients who have received immunotherapeutic drugs such as PD-1 / PD-L1 monoclonal antibody
4. Have received HAIC treatment in the past
5. Severe allergic reaction to other monoclonal antibodies
6. People with known history of central nervous system metastasis or hepatic encephalopathy
7. Patients whose liver tumor burden is greater than 50% of the total liver volume, or who have received liver transplantation in the past
8. Ascites with clinical symptoms, those who need puncture, drainage, or those who have received ascites drainage within the past 3 months, except for those with only a small amount of ascites on imaging but no clinical symptoms
9. Suffer from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
10. Have uncontrolled clinical symptoms or diseases of the heart
11. Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow preventive use of low-dose aspirin and low-molecular-weight heparin
12. Have had significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before randomization
13. Arterial/venous thrombosis events that occurred within 6 months before randomization
14. Known hereditary or acquired bleeding and thrombotic tendency
15. Urine routine test showed urine protein ≥ ++ and confirmed 24-hour urine protein content> 1.0 g
16. Patients who have previously received chemotherapy, hormone therapy, and surgery, after the completion of the treatment (last medication) and less than 4 weeks before the study medication; molecular targeted therapy (including other oral targeted drugs used in clinical trials) is less than 5 drugs from the first study medication Patients whose half-life or adverse events (except alopecia) caused by previous treatment have not recovered to ≤ CTCAE Grade 1
17. The patient has active infection, fever of unknown origin within 7 days before medication ≥38.5℃
18. Patients with congenital or acquired immune deficiencies
19. The patient has suffered from other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ)
20. Patients with bone metastases who received palliative radiotherapy in the 4 weeks before participating in the study >5% of the bone marrow area
21. Live vaccines may be vaccinated during the study period less than 4 weeks before the study medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-10-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (according to mRECIST) | Up to two years
  Time from the first tumor progression or death

SECONDARY OUTCOMES:
Objective response rate (according to mRECIST and RECIST 1.1) | Up to two years
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time (mainly for solid tumors), including complete remission (CR, Complete Response) and partial remission (PR, Partial Response)
Disease control rate (according to mRECIST and RECIST 1.1) | Up to two years
  Refers to the proportion of patients whose tumors have shrunk or been stable for a certain period of time (mainly for solid tumors), including complete remission (CR, Complete Response), partial remission (PR, Partial Response) and stable (SD, Stable Disease)

CONTACTS AND LOCATIONS:
Overall Officials: yue Han, phD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China